CLINICAL TRIAL: NCT06445335
Title: The Prevalence of Non-Alcoholic Fatty Liver Disease in Type 2 Diabetes Mellitus Patients Followed at Ziekenhuis Oost-Limburg, Genk, Belgium
Brief Title: Prevalence of NAFLD in T2DM Patients
Acronym: PAD2ZOL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTU2019009
Record Dates: First submitted 2024-05-21; First posted 2024-06-06 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: NAFLD; T2D; Type 2 Diabetes; Fatty Liver, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FibroScan (Other)
  Interventions: Diagnostic Test: FibroScan

INTERVENTIONS:
Diagnostic Test: FibroScan — Performance of a FibroScan measurement.

SUMMARY:
To determine the prevalence of non-alcoholic fatty liver disease (NAFLD) in patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Having type 2 diabetes mellitus (T2DM)
* Written informed consent obtained

Exclusion Criteria:

* Excessive alcohol use
* Exclusion of other causes of liver disease and secondary causes of steatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of non-alcoholic fatty liver disease (NAFLD) in type 2 diabetes mellitus (T2DM) patients | Baseline
  To determine the prevalence of non-alcoholic fatty liver disease (NAFLD) in type 2 diabetes mellitus (T2DM) patients followed at the department of Endocrinology in Ziekenhuis Oost-Limburg (ZOL), Genk, Belgium by means of FibroScan measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Struyve, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium